CLINICAL TRIAL: NCT05543668
Title: Association of Preoperative Pain With Moderate to Severe Acute Pain After Laparoscopic Cholecystectomy:a Prospective Observational Study.
Brief Title: Association of Preoperative Pain With Moderate to Severe Acute Pain After Laparoscopic Cholecystectomy.
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, BISHAL NEPALI, principal investigator, B.P. Koirala Institute of Health Sciences
Other Study IDs: IRC/2283/022
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Pain, Postoperative
Keywords: postoperative pain, dynamic moderate to severe pain; laprascopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- preexisting preoperative chronic pain: Patients with preexisting preoperative chronic pain (more than 3 months duration).
- preexisting preoperative sub-acute pain: Patients with preexisting preoperative sub-acute pain (less than 3 months duration).
- No pain preoperatively: Patients without preexisting preoperative pain.

SUMMARY:
Despite advancement in perioperative pain management, more than half of the patients still report moderate-severe pain after surgery. Among several risk factors, pre-existing pain has consistently been shown to predict postoperative severe pain.If one can predict the patients who will experience more post-operative pain, then a more aggressive pain management strategy can be adopted perioperatively. This would improve patient satisfaction and prevent poor outcomes such as chronic pain after surgery. Therefore, our primary aim is to find out whether presence of pre-existing preoperative pain would predict moderate-severe acute pain after laparoscopic cholecystectomy. Moreover, we plan to use Patient Reported Outcomes Measurement Information System (PROMIS) scale to assess preoperative pain intensity and pain-related behaviors.

Primary &Secondary Objectives:

Primary objectives To investigate the association between preexisting preoperative pain (more than 3 months duration) and postoperative moderate-severe acute pain after laparoscopic cholecystectomy.

Secondary objectives .1. To investigate the association between preoperative PROMIS(patient reported outcome measurement and information system) domain (PROMIS pain intensity score, PROMIS pain interference score, PROMIS pain behavioural score) and postoperative moderate-severe acute pain after LC.

2. To examine baseline demographic, clinical, psycho-behavioural features and intraoperative factors in relation to dynamic moderate to severe pain after LC.

3. To identify perioperative predictors for acute postsurgical pain. 4. To find out the incidence of shoulder tip pain after LC.

DETAILED DESCRIPTION:
Patients who are 18 years of age or more, of ASA 1, 2 and 3, and scheduled for elective laparoscopic cholecystectomy under general anaesthesia will be enrolled in this prospective observational study. Perioperative anaesthesia management will be standardized for all patients.

Variables such as age, sex, preexisting preoperative pain (chronic or subacute), preoperative PROMIS pain intensity, PROMIS behavior, PROMIS interference, PROMIS depression, PROMIS sleep disturbance, APAIS score, catastrophizing pain score, neuroticism (EPQRS score), preoperative pain sensitivity, an expectation of the postoperative pain and intraoperative surgical variables will be recorded.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing laparoscopic cholecystectomy.

* Age group (more than or equal to 18 years)
* ASA physical status 1, 2 and 3.
* Ability to use NPRS scale, PROMIS scale, pain catastrophizing scale, APAIS, neuroticism EPQRS scale, and to understand and follow simple instructions.

Exclusion Criteria:

All patient with

* Not willing to participate in the study
* Severe Neurological and Psychiatric disorder(eg. dementia)
* Pregnant women
* Acute cholecystitis managed conservatively.
* Cognitive impairments (lack of capacity to provide informed consent)
* Choledocholithiasis
* Features of obstructive jaundice.
* Unable to communicate (eg. Language barrier or deaf)
* Open cholecystectomy or laparoscopic cholecystectomy converted to open cholecystectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 years or more than 18 years of age, ASA PS 1, 2 and 3, scheduled for elective laparoscopic cholecystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of acute moderate to severe postoperative pain. | up to 24 hours postoperatively.
  numerical pain rating scale (NPRS) more than or equal to 4.

SECONDARY OUTCOMES:
incidence of shoulder tip pain. | up to 24 hours postoperatively.
  in 24 hours
Risk factors associated with moderate to severe pain after laparoscopic cholecystectomy | up to 24 hours postoperatively
  demographic, clinical, psycho-behavioural, preoperative and intraoperative variables

CONTACTS AND LOCATIONS:
Overall Officials: Asish Subedi, MD, Study Chair — B.P. Koirala Institute of Health Sciences
Locations (1):
- B.P. Koirala Institute of Health Sciences, Dharān, Province O1, Nepal

IPD SHARING:
Plan to Share IPD: Undecided